CLINICAL TRIAL: NCT00561405
Title: A Motor Learning Based Walking Program Versus Body Weight Supported Treadmill Training in Community Dwelling Adults Within One Year of Stroke Onset: A Randomized Controlled Trial
Brief Title: A Comparison of Two Intensive Walking Training Interventions in Community Dwelling Individuals With History of Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Vince DePaul, Physiotherapist (PT), PhD (candidate), McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06356
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Stroke
Keywords: Stroke; Walking; Motor learning; Skill acquisition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motor Learning Walking Program (Experimental): Motor Learning principles based Walking Program (MLWP) Participants practice variety of real life over ground walking related activities. Order of practice, instructions, guidance and feedback are provided in a manner that facilitates cognitive engagement of learner.
  Interventions: Behavioral: Motor Learning Walking Program
- Body weight supported treadmill training (Active Comparator): Body Weight Supported Treadmill Training. Participants walk on a treadmill while partially supported with an overhead harness system. Mass repetition of the normal gait cycle is encouraged through the support of the harness, the movement of the treadmill, and the assistance of one or two trainers to position limbs and trunk.
  Interventions: Behavioral: Body Weight Supported Treadmill Training

INTERVENTIONS:
Behavioral: Motor Learning Walking Program — Motor Learning principles based Walking Program (MLWP) Participants practice variety of real life over ground walking related activities. Order of practice, instructions, guidance and feedback are provided in a manner that facilitates cognitive engagement of learner. Sessions 45 minutes, 3x per week over 5 weeks for a total of 15 sessions
  Other Names: Task oriented walking training
  Arms: Motor Learning Walking Program
Behavioral: Body Weight Supported Treadmill Training — Participants practice walking on a treadmill while supported with an overhead harness system. Up to 40% body weight support. Target Treadmill speed 2.0 mph. 1 or 2 Trainers (at least one Physical Therapist plus another Physical Therapist or Physiotherapy Assistant) will help guide participants leg, foot and trunk during treatment. Aim is to practice high numbers of repetition of the normal gait cycle on treadmill. Duration of sessions - 20 minutes of treadmill training within a 45 minute session ( 4 sets of 5 minutes of training with 5 minute rests). 3 sessions per week for 5 weeks. Total of 15 sessions.
  Other Names: Treadmill training
  Arms: Body weight supported treadmill training

SUMMARY:
Stroke is a major cause of disability in Canadian adults. Following a stroke, many people have difficulty walking in their home and in the community. The purpose of this study is to compare the effect of two different approaches to walking retraining in people who have had a stroke.

Individuals living in the community who have had recently had a stroke will be asked to participate in this study. Participants will be randomly assigned to one of two five week walking training programs. In one program, individuals will re-learn to walk in a variety of real-life situations. Practice sessions will encourage active problem solving by the participants. The other program will have participants practice walking on a treadmill while some of their body weight is supported by a special harness system. Participants will also be assisted by a physiotherapist to walk in a more normal manner.

Participants' will be assessed at the beginning of the study, after the 5 week training program and again, eight weeks later. The research assistant will assess their ability to walk, their confidence level and the average daily walking activity.

Primary Hypothesis: Individuals assigned to the Motor Learning Walking Program will improve their walking ability from baseline to follow up assessment significantly more than individuals assigned to the Treadmill Training Program.

The results of this study will help physiotherapists plan effective treatment programs for individuals with walking difficulties following stroke. It will also give researchers direction for future studies in the areas of walking retraining and motor skill development post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Stroke onset within previous 12 months
* Age 40 or older
* Able to follow 2 step verbal command (English),
* Able to walk 10 metres without human assistance (may use walking aid)
* Independent community ambulatory prior to stroke
* Community dwelling
* Approval from physician for participation in study

Exclusion Criteria:

* Walking speed greater than 1.0 m/s without walking aid
* Within normal limits on Modified Mini Mental Status test (age and education adjusted)
* Documented global aphasia
* Legal blindness
* Unable to exercise due to the any of the following conditions
* A recent significant change in resting ECG suggesting ischemia
* Recent Myocardial infarction (within 3 months) or other acute cardiac event
* Unstable angina
* Severe SOB at rest or with activities of daily living
* Uncontrolled cardiac arrhythmias causing symptoms
* Severe symptomatic aortic stenosis
* Uncontrolled symptomatic heart failure
* Acute pulmonary embolus or pulmonary infarction
* Acute myocarditis or pericarditis
* Suspected or known dissecting aneurysm
* Acute systemic infection, accompanied by fever, body ache or swollen lymph glands
* Uncontrolled hypertension (systolic > 200 mmHg, diastolic > 110 mmHg )
* Severe peripheral vascular disease with sustained claudication (resulting in limited walking tolerance)
* Severe lower extremity orthopedic problems with severe pain on weight bearing
* Lower extremity amputation that requires prosthesis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-12; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Self selected over ground gait speed - 5 metre walk test | 8 week follow up

SECONDARY OUTCOMES:
Six Minute Walk Test | Post Intervention and 8 week follow up
Self selected over ground gait speed - 5 metre walk test | Post Intervention
Balance related Self Efficacy - Activities-specific Balance Confidence Scale | Post intervention and 8 week follow up
Average Daily Step Count - StepWatch 3 Step Activity Monitor | Post Intervention and 8 Week Follow up
Dynamic Balance - Functional Balance Test | Baseline, Post-intervention and 8 week Follow-up
  Over a 9 m track - participants are required to perform 5 balance and walking related tasks. Participants are required to 1) rise from a chair, walk 3 m, 2) step up and down an 8 inch step, walk 3 m, 3) bend down to pick up and return a 2.5 kilo weight off floor, walk 3 m to marked spot on the floor, 4) turn 180 degrees and walk 9 m back to the chair, 5. sit back down in the chair.
  Each task is scored on a 4 point scale (total score of out 20) Participants are timed on how long it takes them to perform the entire circuit.
Life Space Questionnaire | Baseline, Post-intervention, and at 8 week follow up
  Self-report measure of mobility partipation.
Number of trainers required per treatment session | Documented at every treatment session for both experimental and active comparison interventions.
Patient Specific Functional Scale | Baseline, Post-intervention, Follow-up (8weeks)
  In this measure, participants are asked to identify 3 walking related functional activities that they currently have some difficulty performing and would like to improve with treatment. For each activity, the participant rates their current ability to perform the task on a numeric rating scale of 0 to 10.
  At Post-intervention and Follow-up, participants re-rate their current ability on the same activites (without seeing their previous score).
Rating of Walking functional level - Modified Functional Walking Categories | Baseline, Post-intervention, Follow-up (8 weeks)
Adverse event - Self-report of a fall(s) since baseline assessment | Post Intervention Assessment
  Participants will be asked whether or not they have had a fall since baseline assessment. Details of the fall(s) will be recorded. Fall report based on participant recall - no other tools (e.g. diary) will be used.
Adverse event - Falls (yes or no) | Follow - up - 8 weeks after post-intervention assessment
  Participant asked to report whether or not they had a fall since Post Intervention assessment. Details of the fall will be provided.
  Based on participant recall - no other tools for falls recording will be used (ie. will not be using falls diary)
Serious adverse events - ie. new stroke, myocardial infarction, overnight hospital admission, death | Post-intervention, Follow up (8 weeks)
  Serious adverse events will be based on participant or caregiver report, and confirmed with primary care physician as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent G DePaul, PhD (c), Principal Investigator — McMaster University, Hamilton, ON, Canada
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] DePaul VG, Wishart LR, Richardson J, Lee TD, Thabane L. Varied overground walking-task practice versus body-weight-supported treadmill training in ambulatory adults within one year of stroke: a randomized controlled trial protocol. BMC Neurol. 2011 Oct 21;11:129. doi: 10.1186/1471-2377-11-129. PMID 22018267